CLINICAL TRIAL: NCT02539758
Title: The Effect of Ocular Massage on the Management of Elevated Intraocular Pressure After Acute Angle Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lv Yingjuan (Other)
Responsible Party: Sponsor-Investigator, Lv Yingjuan, department of ophthamology, Tianjin Medical University Eye Hospital
Organization: Tianjin Medical University Eye Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: tjykdxykyy2
Record Dates: First submitted 2015-08-08; First posted 2015-09-03 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-08

CONDITIONS: Intraocular Pressure
Keywords: acute angle closure; ocular massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ocular massage (Experimental): over the closed eyelids with moderate massage strength for 15 minutes. The compression of the globe was given with finger, and press for 2 seconds, then by a 2 seconds release, with a frequency of 15 presses/minute.We observed changes of anterior chamber depth before and after ocular massage by LenstarLS900,and changes of intraocular pressure before and after ocular massage by Goldmann tonometer
  Interventions: Other: ocular massage; Device: LenstarLS900; Device: Goldmann tonometer

INTERVENTIONS:
Other: ocular massage — ocular massage could be applied over the globe over the closed eyelids with moderate massage strength for 15 minutes. The compression of the globe was given with finger, and press for 2 seconds, then by a 2 seconds release, with a frequency of 15 presses/minute.
Device: LenstarLS900 — observed changes of anterior chamber depth before and after ocular massage by LenstarLS900
Device: Goldmann tonometer — observed changes of intraocular pressure before and after ocular massage by Goldmann tonometer

SUMMARY:
Lowering intraocular pressure remains the mainstay of therapy in the management of glaucoma. The effect of ocular massage on intraocular pressure in patients with acute primary angle closure was the important thing.This was a prospective study, in which 20 eyes from 20 patients had acute angle closure. When they went to the hospital, ocular massage was performed without any medication. Intraocular pressure was detected by Goldmann tonometer, and Lenstar LS900 optical biometry observed changes of anterior chamber depth before and after ocular massage. Anterior chamber depth, anterior chamber angle and ciliary body were observed by Ultrasound biomicroscopy after massage, and anterior chamber angle was also checked by gonioscope after massage.

DETAILED DESCRIPTION:
Background: Primary angle closure glaucoma is still the most common type in Asia. Lowering intraocular pressure remains the mainstay of therapy in the management of glaucoma, since it has been shown to be effective in reducing optic nerve damage and loss of vision. The objective of this study was to evaluate to assess the effect of ocular massage on intraocular pressure in patients with acute primary angle closure.

Methods : This was a prospective study, in which 20 eyes from 20 patients had acute angle closure. When they went to the hospital, ocular massage was performed without any medication. Intraocular pressure was detected by Goldmann tonometer, and Lenstar LS900 optical biometry (Lenstar LS900) observed changes of anterior chamber depth before and after ocular massage. Anterior chamber depth, anterior chamber angle and ciliary body were observed by Ultrasound biomicroscopy (after massage, and anterior chamber angle was also checked by gonioscope after massage.

ELIGIBILITY:
Inclusion Criteria:

* All of them had documented evidence of acute angle closure.

Exclusion Criteria:

-

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
observed changes of anterior chamber depth before and after ocular massage | before ocular massage and 15 minutes after massage

SECONDARY OUTCOMES:
observed changes of intraocular pressure before and after ocular massage | before ocular massage and 15 minutes after massage

CONTACTS AND LOCATIONS:
Overall Officials: yingjuan Lv, Principal Investigator — Tianjin Medical University Eye Hospital
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality, China